CLINICAL TRIAL: NCT04288570
Title: Punch vs. Drill Tunnel Use for Anchor Tunnel Creation and Correlation With Post-operative Pain
Acronym: Punch/Drill
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Matt Smith (Other)
Responsible Party: Sponsor-Investigator, Matt Smith, ASSOCIATE PROFESSOR OF CLINICAL, MOI OUTPATIENT MEDICAL DIRECTOR, Orthopaedic Surgery, University of Missouri-Columbia
Organization: University of Missouri-Columbia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019842
Record Dates: First submitted 2020-02-20; First posted 2020-02-28 (Actual); Results first posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Rotator Cuff Tears
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bone socket formation with a punch (Active Comparator): suture anchor socket creation with punch
  Interventions: Procedure: suture anchor socket creation with punch
- Bone socket formation with a drill (Active Comparator): suture anchor socket creation with drill
  Interventions: Procedure: suture anchor socket creation with drill

INTERVENTIONS:
Procedure: suture anchor socket creation with punch — suture anchor socket creation with punch
  Arms: Bone socket formation with a punch
Procedure: suture anchor socket creation with drill — suture anchor socket creation with drill
  Arms: Bone socket formation with a drill

SUMMARY:
To determine if different techniques used in the creation of suture anchor socket creation can influence post-op pain following rotator cuff repair.

ELIGIBILITY:
Inclusion Criteria:

a. Patient's aged 18-80 years old with diagnosis of rotator cuff tear having failed non-operative management and being indicated for surgical intervention with use of suture anchors.

Exclusion Criteria:

1. Glenohumeral arthrosis
2. Previous shoulder surgery
3. Psychiatric diseasesMRI
4. Rheumatologic diseases
5. Fibromyalgia
6. Spine diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Smith, Principal Investigator — University of Missouri Health System, Department of Orthopaedic Surgery
Locations (1):
- University of Missouri, Columbia, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bone Socket Formation With a Punch | Bone Socket Formation With a Drill
Started | 21 | 22
Completed | 21 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bone Socket Formation With a Punch | Bone Socket Formation With a Drill | Total
Number analyzed (Participants) | 21 | 22 | 43
Age, Continuous [Mean (Full Range); unit: years] | 61.4 [36 to 72] | 59.3 [43 to 80] | 60.3 [36 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 12 | 19
  Male | 14 | 10 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 21 | 18 | 39
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) - Physical Function Short Form
Description: The PROMIS Physical Function Short Form uses T-scores (Mean = 50, SD = 10), where higher scores indicate better physical function. Responses use a Likert scale: 1 = "Unable to do," 2 = "With much difficulty," 3 = "With some difficulty," 4 = "With a little difficulty," 5 = "Without any difficulty." Raw scores are summed and converted to T-scores. 50 = average function, 60 = 1 SD above (better), 40 = 1 SD below (worse).
Time Frame: Preop, 2 Weeks, 6 Weeks, 3 Months, 6 Months
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Bone Socket Formation With a Punch | Bone Socket Formation With a Drill
Number analyzed (Participants) | 21 | 22
T-Score
  Preop | 41.51 (2.22) | 40.54 (2.24)
  2 Weeks | 36.81 (2.42) | 32.16 (2.58)
  6 Weeks | 42.74 (2.42) | 37.90 (2.52)
  3 Months | 44.41 (2.23) | 42.22 (2.24)
  6 Months | 46.90 (2.52) | 46.31 (2.31)

2. Primary Outcome: Single Assessment Numeric Evaluation (SANE)
Description: The Single Assessment Numeric Evaluation (SANE) is a simple, one-question patient-reported outcome measure. A SANE score requires the patient to rate their knee function on a scale of 0 to 100% with 100% being normal.
Time Frame: Preop, 2 Weeks, 6 Weeks, 3 Months, 6 Months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bone Socket Formation With a Punch | Bone Socket Formation With a Drill
Number analyzed (Participants) | 21 | 22
score on a scale
  PreOp | 35.86 (17.22) | 32.14 (21.76)
  2 Weeks | 22.0 (22.67) | 17.06 (22.10)
  6 Weeks | 35 (29.53) | 22.5 (14.62)
  3 Months | 38.83 (25.14) | 47.2 (24.27)
  6 Months | 68.36 (31.63) | 76.23 (20.67)

3. Primary Outcome: Visual Analogue Scale
Description: Patient Reported Outcome Measure - pain Scale: 0-10. 0 being no pain and 10 being unbearable pain
Time Frame: Preop, 2 Weeks, 6 Weeks, 3 Months, 6 Months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bone Socket Formation With a Punch | Bone Socket Formation With a Drill
Number analyzed (Participants) | 21 | 22
score on a scale
  Preop | 4.86 (2.01) | 4.95 (2.48)
  2 Weeks | 1.14 (1.46) | 3.56 (2.83)
  6 Weeks | 1.78 (1.62) | 2.11 (2.51)
  3 Months | 2.06 (1.84) | 2.33 (1.96)
  6 Months | 2.64 (2.42) | 2.54 (2.50)

4. Primary Outcome: PROMIS - Pain Interference
Description: The PROMIS Pain Interference Short Form uses T-scores (Mean = 50, SD = 10), where higher scores indicate greater pain interference. Responses use a Likert scale: 1 = "Not at all," 2 = "A little bit," 3 = "Somewhat," 4 = "Quite a bit," 5 = "Very much." Raw scores are summed and converted to T-scores. 50 = average pain interference, 60 = 1 SD above (worse), 40 = 1 SD below (better).
Time Frame: Preop, 2 Weeks, 6 Weeks, 3 Months, 6 Months
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Bone Socket Formation With a Punch | Bone Socket Formation With a Drill
Number analyzed (Participants) | 21 | 22
T-Score
  Preop | 62.23 (1.74) | 63.11 (1.84)
  2 Weeks | 54.76 (1.95) | 61.66 (2.43)
  6 Weeks | 55.02 (1.98) | 58.52 (2.58)
  3 Months | 55.51 (1.93) | 56.83 (2.03)
  6 Months | 54.20 (3.0) | 54.27 (2.55)

5. Secondary Outcome: Magnetic Resonance Imaging (MRI) of the Shoulder
Description: MRI of the shoulder of the first 5 patients in each group will be obtained at 2 weeks post-op for evaluation of bone marrow lesion in the proximal humerus. Bone marrow lesion size measured in mm2 on a calibrated MR image from 0 (no lesion, better) to 180 (large lesion, worse)
Time Frame: 2 weeks
Population: The analysis population include all participants that completed the MRI at the 2 week post-op evaluation.
Measure: Mean (Full Range); unit: mm^2
Arm/Group | Bone Socket Formation With a Punch | Bone Socket Formation With a Drill
Number analyzed (Participants) | 5 | 4
mm^2 | 20.4 [11.8 to 29.4] | 21.7 [12.7 to 33.3]

ADVERSE EVENTS:
Time Frame: 6 Months
Arm/Group | Bone Socket Formation With a Punch | Bone Socket Formation With a Drill
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/22
Other Adverse Events (participants affected / at risk) | 0/21 | 0/22

LIMITATIONS AND CAVEATS:
A limitation of our study was that the surgeon was not blinded to the intervention given that surgical technique was the variable in question for the study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2020-02-24): https://cdn.clinicaltrials.gov/large-docs/70/NCT04288570/Prot_000.pdf